CLINICAL TRIAL: NCT00002153
Title: Topical Use of 4,4'-Dihydroxybenzophenone-2,4-Dinitrophenylhydrazone (A-007) in the Treatment of Advanced Malignancies Including Kaposi's Sarcoma and Lymphoproliferative Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DEKK-TEC, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 247A; DTI-006
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-05

CONDITIONS: Sarcoma, Kaposi; HIV Infections; Lymphoproliferative Disorders
Keywords: Skin Neoplasms; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Antineoplastic Agents
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Lymphoproliferative Disorders; Skin Neoplasms; Acquired Immunodeficiency Syndrome | interventions — 4,4'-dihydroxybenzophenone-2,4-dinitrophenylhydrazone

INTERVENTIONS:
Drug: A-007

SUMMARY:
To evaluate topical A-007 in patients with advanced malignancies including Kaposi's sarcoma and lymphoproliferative disorders.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Maintenance antihormones, hormones, and glucocorticoids.

Patients must have:

* Histologically proven metastatic cancer including Kaposi's sarcoma and lymphoproliferative disorders to the skin or cutaneous sites. NOTE:
* Primary basal or squamous cell cancer of the skin is allowed.
* Failed both primary and secondary chemotherapy and/or immunotherapy protocols.
* Measurable skin or cutaneous lesions. 4 Life expectancy of at least 20 weeks.

Prior Medication:

Required:

* Prior therapy for cutaneous lesions from Kaposi's sarcoma or lymphoproliferative disorders.

Allowed:

* Prior maintenance steroids and hormone/antihormone therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active infections other than medically stable HIV infection.
* Active congestive heart failure, any persistent arrhythmia or transient serious arrhythmia (ventricular tachycardia, sinoatrial arrest, etc.), or progressive cardiomyopathy.
* Unstable blood pressure.
* Seizures or other CNS disorders.
* Severe unstable diabetes mellitus.
* Coagulopathies.
* Thrombotic disease.
* Any other medical conditions that would prevent completion of study or produce significant risk to patient.

Concurrent Medication:

Excluded:

* Concomitant chemotherapy or immunotherapy.
* Ongoing corticosteroid therapy (unless maintenance).

Patients with the following prior conditions are excluded:

* History of active cardiopulmonary or respiratory disease.
* History of sun hypersensitivity and photosensitive dermatoses.
* History of allergy or hypersensitivity to cosmetics, toiletries, or other dermatological products.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25

CONTACTS AND LOCATIONS:
Locations (1):
- DEKK - TEC Inc, New Orleans, Louisiana, United States